CLINICAL TRIAL: NCT03676699
Title: Lung Ultrasound as an Evolving Tool in Detection of Extravascular Lung Water in Septic Cancer Patients.
Brief Title: Lung Ultrasound in Detection of Extravascular Lung Water in Septic Patients.
Status: Completed | Type: Observational
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ehab Hanafy Shaker, lecturer of anesthesia ,critical care and pain medicine, National Cancer Institute, Egypt
Other Study IDs: Ehab-Walaa.Ultrasound
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Ultrasound Therapy; Complications
Keywords: Extravascular lung water, inferior vena cava collapsibility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound chest — Ultrasound detection of extravascular lung water

SUMMARY:
Sepsis is a common serious problem in surgical critical care units.Septic shock can be a consequence of severe sepsis with high mortality rate, in which there is major disturbance on the cellular, metabolic and circulatory levels.Patients who suffer from malignancy or under chemotherapeutic treatment are at higher risk of sepsis.Postoperative cancer patients carry both the risk of underlying malignancy with superimposed risk of major surgical procedure.]. Monitoring effective fluid resuscitation and patient's hemodynamic status is achieved through different techniques mainly by measuring central venous pressure (CVP), pulmonary artery occlusion pressure (PAOP) and transpulmonary thermodilution along with chest radiography analysis .This study aims to investigate the correlation between lung ultrasound and IVC collapsibility index in assessment of fluid responsiveness in cancer patients with septic shock.

DETAILED DESCRIPTION:
Sepsis is a common serious problem in surgical critical care units.Septic shock can be a consequence of severe sepsis with high mortality rate, in which there is major disturbance on the cellular, metabolic and circulatory levels . Patients who suffer from malignancy or under chemotherapeutic treatment are at higher risk of sepsis.Postoperative cancer patients carry both the risk of underlying malignancy with superimposed risk of major surgical procedure.Upon recognition of septic shock, management should start promptly, aiming at effective restoration of the intravascular volume, identification, control of source of infection and starting empiric intravenous antimicrobials. This is a common problem in critically ill patients especially in presence of sepsis. Monitoring effective fluid resuscitation and patient's hemodynamic status is achieved through different techniques mainly by measuring central venous pressure (CVP), pulmonary artery occlusion pressure (PAOP) and transpulmonary thermodilution along with chest radiography analysis.Recently lung ultrasound evolved as a novel tool for assessment of extravascular lung water (EVLW) and lung congestion. It is a bed side noninvasive assessment tool. EVLW accumulation is diagnosed through interpretation of B-Lines which are echoic Vertical, comet-tail-like lines extending from the pleura line to the screen edge without fading .The normal lung pattern of no-echo signal or black lung, changes into black and white pattern with lung congestion, then into white lung pattern with alveolar pulmonary edema .This study aims to investigate the correlation between lung ultrasound and IVC collapsibility index in assessment of fluid responsiveness in cancer patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between (18 - 65) years.
* Diagnosed with severe sepsis or septic shock according to the third international consensus definition (sepsis-3).
* All of them underwent major abdominal oncologic surgeries.

Exclusion Criteria:

* ASA III and IV patients.
* Patients with BMI>35.
* Patients who suffered from chronic lung disease.
* History of cardiac or renal problems.
* Patients with lung cancer or pulmonary metastases.
* Patients with inserted chest tubes.
* Presence of subcutaneous emphysema.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients meeting the inclusion criteria with severe sepsis and septic shock admitted to the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Detection of B-lines | 12 hours follow up
  The number of B lines was scanned and a quadrant was considered to be positive when 3 or more B-Lines were recorded. A patient was defined to have positive B-lines (when 3 or more B-Lines are recorded in 3 or more quadrants).

CONTACTS AND LOCATIONS:
Overall Officials: Ehab H Shaker, MD, Principal Investigator — National Cancer Institute- Cairo University
Locations (1):
- Department of Anesthesia and Pain medicine.National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
after finishing the submission ,we planned to share the results and conclusion for further benefits.

REFERENCES:
- See also: Lung ultrasonography for the assessment of rapid extravascular water variation: evidence from hemodialysis patients. — https://www.ncbi.nlm.nih.gov/pubmed/21590437